CLINICAL TRIAL: NCT00692315
Title: Efficacy of Methylcobalamin and Folinic Acid Treatment on Glutathione Redox Status and Core Behavior in Children With Autism
Brief Title: Treating Oxidative Stress in Children With Autism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arkansas Children's Hospital Research Institute (Other)
Responsible Party: S. Jill James, Arkansas Children's Hospital Research Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 28839
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Autistic Disorder
Keywords: glutathione; methionine; folinic acid; redox; oxidative stress; behavior
MeSH Terms: conditions — Autistic Disorder; Behavior | interventions — mecobalamin; Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methyl B12 (Experimental): Subcutaneous injection of 75 micrograms/Kg
  Interventions: Drug: Methylcobalamin (methylB12)
- Folinic Acid (Experimental): 400 micrograms orally twice a day
  Interventions: Drug: Methylcobalamin (methylB12)

INTERVENTIONS:
Drug: Methylcobalamin (methylB12) — 75 ug/Kg methylB12 every 3 days by subcutaneous injection
  Other Names: Vitamin B12

SUMMARY:
An open label trial was undertaken in 40 autistic children to determine whether treatment with metabolic precursors methylcobalamin and folinic acid would improve plasma biomarkers of oxidative stress and measures of core behavior using the Vineland Adaptive Behavior Scales (VABS). Metabolites involved in methionine and glutathione synthesis and VABS behavior scores were measured before and after a three month intervention period.

The results indicated that pre-treatment metabolites in autistic children were significantly different from values in age-matched control children. The three month intervention resulted in significant increases in cysteine, cysteinylglycine, and glutathione (GSH, p < 0.001). The oxidized disulfide form of glutathione (GSSG) was decreased (p < 0.008) and the glutathione redox ratio (GSH/GSSG) was increased after treatment (p < 0.001). Although significantly improved, these metabolites remained below control levels after intervention (p > 0.01). Similarly, increases in VABS composite score and sub-scores for Socialization, Communication, and Daily Living Skills increased after treatment (p < 0.007) but also remained below standard scores.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Autistic Disorder by DSM-IV 299.0 or CARS score >30

Exclusion Criteria:

* Primary genetic disease with co-morbid autism
* frequent seizures
* recent surgery
* active infection with fever
* high dose vitamin/mineral supplements
* severe gastrointestinal symptoms

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2006-09; Primary Completion 2007-06 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Glutathione redox status (GSH/GSSG) | 3 months
  HPLC analysis

SECONDARY OUTCOMES:
Vineland Adaptive Behavior Scales | 3 months
  Behavior measure

CONTACTS AND LOCATIONS:
Overall Officials: S. Jill James, PhD, Principal Investigator — University of Arkansas
Locations (1):
- Arkansas Children's Hospital Research Institute, Little Rock, Arkansas, United States

REFERENCES:
- [Derived] James SJ, Melnyk S, Fuchs G, Reid T, Jernigan S, Pavliv O, Hubanks A, Gaylor DW. Efficacy of methylcobalamin and folinic acid treatment on glutathione redox status in children with autism. Am J Clin Nutr. 2009 Jan;89(1):425-30. doi: 10.3945/ajcn.2008.26615. Epub 2008 Dec 3. PMID 19056591